CLINICAL TRIAL: NCT04789421
Title: Multicenter, Randomised Study of the Impact of Advanced, Non-invasive Diagnostic Instrumentation for Early Cutaneous Tumor Diagnosis, Clinical-therapeutic Pathways and an Economic-management Perspective
Brief Title: Advanced Non-invasive Diagnostics for Early Cutaneous Tumor Diagnosis, Clinical-therapeutic and Economic Management
Acronym: NET-DAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Pellacani Giovanni, Professor of Dermatology, Azienda Ospedaliero-Universitaria di Modena
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: NET-2011-02347213; 3844/C.E. (Other: University-Hospital of Modena Provincial Ethics Committee)
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Cutaneous Melanoma
Keywords: diagnostic accuracy; number needed to excise; reflectance confocal microscopy; histopathology; dermoscopy; early diagnosis
MeSH Terms: conditions — Melanoma; Disease | interventions — Dermoscopy

STUDY DESIGN:
Intervention Model Description: A two-arm prospective, multi-center study of the triage of patients with equivocal skin lesions suspicious for melanoma, compared with the standard of care (i.e. clinical and dermoscopic examination). A 1:1 randomization into the interventional or control arms occurred at the time of enrolment. Arm 1 (interventional) included lesions that were evaluated with RCM with management decisions taken according with overall information (2 possible outcomes: excision or digital monitoring. Arm 2 (control) included lesions that were not evaluated with RCM, with management decisions taken according to clinical and dermoscopy evaluations only (2 possible outcomes: excision or follow-up).
Who Masked: Care Provider
Masking Description: Randomisation of patients to Arm 1 (with RCM evaluation) or Arm 2 (without RCM evaluations) was performed following clinical and dermoscopy evaluation, and was only revealed to the clinician at presentation of RCM evaluation request.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm 1 (interventional) (Active Comparator): Patients with equivocal skin lesions suspicious for melanoma, randomised to adjunctive RCM evaluation, following clinical and dermoscopy evaluation.
  Interventions: Device: Clinical, dermoscopy and Reflective confocal microscopy evaluations
- Arm 2 (control) (Placebo Comparator): Patients with equivocal skin lesions suspicious for melanoma, randomised to clinical and dermoscopy evaluation only; adjunctive RCM evaluation refused.
  Interventions: Device: Clinical, dermoscopy evaluations

INTERVENTIONS:
Device: Clinical, dermoscopy and Reflective confocal microscopy evaluations — Adjunctive reflective confocal microscopy to dermoscopy and clinical dermatological evaluation.
  Arms: Arm 1 (interventional)
Device: Clinical, dermoscopy evaluations — Dermoscopy and clinical dermatological evaluation only
  Arms: Arm 2 (control)

SUMMARY:
The incidence of cutaneous melanoma (MM) is increasing worldwide. The best therapeutical solution for MM is early diagnosis and efforts over the last 50 years have been directed towards early and precise diagnoses.

Dermoscopy has improved diagnostic accuracy compared to the naked eye, but is limited by an associated higher number of unnecessary excisions. Reflectance confocal microscopy (RCM) is a novel technique enabling in vivo examination of the skin at cellular-level resolution, with excellent diagnostic accuracy.

This study hypothesis is that the systematic application of RCM in the triage and management of patients suspicious for skin cancer, may improve diagnostic accuracy and reduce the number of unnecessary biopsy. Reducing the burden of unnecessary surgery excisions should benefit the health system, both in saving surgical and pathology procedural associated costs and reducing the overwhelming waiting lists for excisions and consequent risk for delayed diagnoses.

ELIGIBILITY:
Inclusion Criteria:

- Patient's with at least 1 unequivocal lesion following standard of care (clinical and dermoscopy evaluations), >= 18 years old

Exclusion Criteria:

* (i) the presence of an unequivocal aspect of melanoma or of any other malignant skin cancer,
* (ii) lesion located on a skin area where reflectance confocal microscopy cannot be performed (for example: skin folds, mucosa, etc.),
* (iii) lesion larger than 2 cm in its largest diameter
* (iv) lesion where RCM examination is hampered for over the 30% of its surface (for example, for presence of crusting, oozing, erosion, ulceration, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3248 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Number needed to excise (NNE) | 03/2016 - 02/2020
  Measure the number of lesions needed to excise for a cutaneous melanoma diagnosis
Early diagnosis | 03/2016 - 02/2020
  Measure the breslow index of excised lesions
RCM diagnostic sensibility and sensitivity | 03/2016 - 02/2020
  Diagnostic sensibility of RCM in identifying cutaneous melanoma among equivocal lesions suspicious for melanoma (without clear demoscopy criteria for melanoma)

SECONDARY OUTCOMES:
Head and neck pigmented lesions | 03/2016 - 02/2020
  Diagnostic accuracy of pigmented head and neck lesions where differential diagnosis is difficult to achieve and improper treatments (cryotherapy, laser, radiofrequency).
Diagnostic accuracy of non melanoma skin cancer | 03/2016 - 02/2020
  Pre-and intra-operative imaging for surgical margins

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Pellacani, MD, Principal Investigator — Azienda Ospedaliera Modena

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a sharing platform
Supporting Information: Study Protocol
Time Frame: Data will be available in 2021

REFERENCES:
- [Derived] Longo C, Guida S, Mirra M, Pampena R, Ciardo S, Bassoli S, Casari A, Rongioletti F, Spadafora M, Chester J, Kaleci S, Lai M, Magi S, Mazzoni L, Farnetani F, Stanganelli I, Pellacani G. Dermatoscopy and reflectance confocal microscopy for basal cell carcinoma diagnosis and diagnosis prediction score: A prospective and multicenter study on 1005 lesions. J Am Acad Dermatol. 2024 May;90(5):994-1001. doi: 10.1016/j.jaad.2024.01.035. Epub 2024 Jan 30. PMID 38296197
- [Derived] Pellacani G, Farnetani F, Ciardo S, Chester J, Kaleci S, Mazzoni L, Bassoli S, Casari A, Pampena R, Mirra M, Lai M, Magi S, Mandel VD, Di Matteo S, Colombo GL, Stanganelli I, Longo C. Effect of Reflectance Confocal Microscopy for Suspect Lesions on Diagnostic Accuracy in Melanoma: A Randomized Clinical Trial. JAMA Dermatol. 2022 Jul 1;158(7):754-761. doi: 10.1001/jamadermatol.2022.1570. PMID 35648432